CLINICAL TRIAL: NCT03584399
Title: Prospective Incidence of Persistent Inflammatory, Immunosuppressed, Catabolic Syndrome in the Critically Ill Pediatric Population
Brief Title: Prospective Evaluation of the Incidence of PICS
Acronym: ProsPICS
Status: Terminated | Type: Observational
Why Stopped: lack of enrollment
Sponsor: Indiana University (Other)
Collaborators: American Society for Parenteral and Enteral Nutrition (Other)
Responsible Party: Principal Investigator, Courtney Rowan, Assistant Professor Pediatrics, Indiana University
Other Study IDs: 1802247905
Record Dates: First submitted 2018-06-04; First posted 2018-07-12 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Metabolism and Nutrition Disorder
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In addition to CRP and TLC, which will be collected at 14 days (± 1 day) of PICU admission , an additional blood samples will be collected at these time points to be frozen for further analysis. At the time of blood collection, an additional 5 mL of blood will be collected, processed, and stored at -80 degree Celsius. Once desired time-points are identified and further funding obtained, samples will be processed in batches to evaluate biochemical markers of inflammation. This will be performed using The Inflammatory Cytokine Human Magnetic 5-Plex Panel for the Luminex™ platform. This will quantify GM-CSF, IL-1β, IL-6, IL-8 and TNF-α in serum samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PICS in critically ill pediatric population — Collection of additional blood sample from those subjects meeting criteria for the study.

SUMMARY:
Advances in modern medicine and critical care interventions have greatly impacted survival of critically ill patients, but these interventions are not without consequences. Although patients may now survive the initial critical illness, these patients may not recover to their pre-illness baseline state of health. Recent data in both the critically ill adult and neonatal patients who survive sepsis or surgical events have been shown to progress to persistent inflammatory, immunosuppressed, catabolic syndrome (PICS). This was first identified in adult trauma patients, and more recently was defined in critically ill neonates. To date, there are no published reports of PICS in the critically ill pediatric population. Our long-term goal is to understand PICS in the pediatric population and how early medical and nutritional interventions may impact overall morbidity and survival. To achieve this goal first PICS must first be characterized in the pediatric population. The hypothesis is that PICS occurs in pediatric patients and is associated with increased time to return to a baseline functional life post-injury or illness. The hypothesis will be tested by pursuing the following specific aims. Specific Aim 1: To determine the incidence of PICS in the pediatric population and associate the diagnosis of PICS to survival and time to return to baseline functional life and Specific Aim 2: To determine if early increased inflammatory and immunosuppressive markers are associated with the development of PICS and increased morbidity and mortality. These aims will be accomplished by conducting a prospective single-center observational pilot study to enroll pediatric patients with an anticipated pediatric intensive care unit (PICU) stay greater than 14 days. Through these two aims, the investigators anticipate that this research will provide an explanation into the interplay of inflammation, immunosuppression, and catabolism in critically ill children, which is imperative to the development of early therapeutic and nutritional interventions that can reduce morbidity and mortality associated with critical illness.

DETAILED DESCRIPTION:
The long-term goal of this study is to understand PICS in the pediatric population and how early medical and nutritional interventions may impact overall morbidity and survival, but first PICS must be characterized in the pediatric population. The hypothesize is that PICS occurs in pediatric critically ill patients and is associated with increased time to return to a baseline functional life post-injury or illness.

Enrollment/Randomization This is a prospective observational study with no randomization. The patients will be approached between PICU stay days 9-12 for consent. Labs will be drawn between PICU stay days 12-16 with a preference for PICU day 14, however, labs will be drawn in accordance with the standard of care labs to avoid additional draws.

Study Procedures

Specific Aim 1: To determine the incidence of PICS in the pediatric population and associate the diagnosis of PICS to survival and time to return to baseline functional life.

In order to determine the incidence of PICS in PICU patients, a prospective single-center study will be conducted of all critically ill pediatric patients admitted to PICU at Riley Hospital for Children at Indiana University Health, Indianapolis, IN. Patients will be included if they have an anticipated stay of >14 days in the PICU. Patients will be excluded from this study if they have are maintained on chronic mechanical ventilation, have a known chronic inflammatory disease process, or are diagnosed with failure to thrive or malnutrition upon admission to the PICU.

Data to be collected will include demographic data, nutrition data (weight, protein/non-protein calories received, type of nutrition and prescribed goal nutrition by a dietician), severity of illness, length of stay in the PICU and hospital. Existing routine labs from admission and PICU stay including blood counts, electrolytes and nutrition labs will be collected. At 14 days (± 1 day) the patient will be approached for inclusion into the study. At that time, routine labs to check for inflammation and nutritional status such as CRP, total lymphocyte count, albumin, prealbumin, and retinol binding protein will be collected Diagnosis of PICS will be determined when a patient has been admitted to the PICU for >14 days and has signs of both inflammation (CRP >15mg/L) and immunosuppression (total lymphocyte count < 0.80×109/L), as well as catabolism (Serum albumin < 3.0g/dL, Prealbumin <10mg/dL, Retinol binding protein <10μg/dL, and weight loss >10% or body mass index <18 during hospitalization).

Data Management:

Data will be entered and stored in in a de-identified/HIPAA compliant manner using a password protected web-based database that has securities to protect confidentiality and data integrity. The database will be constructed in REDCap.

Data Analysis Plan:

Clinical risk factors will be summarized and distributions examined. Relationships between the variables and the development of PICS will be explored using plots, correlation coefficients, and contingency tables. The association between clinical variables, including nutritional interventions, and PICS will then be analyzed with logistic regression. Both univariate and multivariate analyses will be conducted. The significance threshold p-value is set at 0.05.

Specific Aim 2: To determine if early increased inflammatory and immunosuppressive markers are associated with the development of PICS and increased morbidity and mortality.

Sample management and processing:

In addition to CRP and TLC, which will be collected at 14 days (± 1 day) of PICU admission , additional blood samples will be collected at these time points to be frozen for further analysis. At the time of blood collection, an additional 5 mL of blood will be collected, processed, and stored at -80 degree Celsius. Once desired time-points are identified and further funding obtained, samples will be processed in batches to evaluate biochemical markers of inflammation. This will be performed using The Inflammatory Cytokine Human Magnetic 5-Plex Panel for the Luminex™ platform. This will quantify GM-CSF, IL-1β, IL-6, IL-8 and TNF-α in serum samples.

The expected outcomes will focus on characterizing PICS in the pediatric population and identifying early inflammatory markers that may correlate with the development of PICS and subsequently increased morbidity associated with critical illness. The results are expected to have a positive impact by filling a key gap in the understanding of the mechanism of PICS in critically ill children. This research will provide insight into the interplay of inflammation, immunosuppression, and catabolism in critically ill children, which is imperative to the development of early therapeutic and nutritional interventions that can reduce morbidity and mortality associated with critical illness.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are < or = to 18 years of age and have an anticipated length of PICU stay of > or = to 14 days from June 1, 2018 through January 31, 2019

Exclusion Criteria:

* Chronic mechanical ventilation, Known chronic inflammatory disease process, or Diagnosed with failure to thrive or malnutrition upon admission to the PICU

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects will be admitted the to pediatric intensive care unit of Riley Hospital for Children.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of PICS in the pediatric critical care population | July 1, 2018 to June 30, 2019
  Diagnosis of PICS will be determined when a patient has been admitted to the PICU for >14 days and has signs of both inflammation (CRP >15mg/L) and immunosuppression (total lymphocyte count < 0.80×109/L), as well as catabolism (Serum albumin < 3.0g/dL, Prealbumin <10mg/dL, Retinol binding protein <10μg/dL, and weight loss >10% or body mass index <18 during hospitalization).

SECONDARY OUTCOMES:
Mortality | July 1, 2018 to June 30 2019
  Death in the ICU associated with PICS

CONTACTS AND LOCATIONS:
Overall Officials: Courtney M Rowan, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Data will be entered and stored in in a de-identified/HIPAA compliant manner using a password protected web-based database that has securities to protect confidentiality and data integrity. The database will be constructed in REDCap.

REFERENCES:
- [Background] Epstein D, Brill JE. A history of pediatric critical care medicine. Pediatr Res. 2005 Nov;58(5):987-96. doi: 10.1203/01.PDR.0000182822.16263.3D. Epub 2005 Sep 23. PMID 16183804
- [Background] Marshall JC. Critical illness is an iatrogenic disorder. Crit Care Med. 2010 Oct;38(10 Suppl):S582-9. doi: 10.1097/CCM.0b013e3181f2002a. PMID 21164401
- [Background] Gentile LF, Cuenca AG, Efron PA, Ang D, Bihorac A, McKinley BA, Moldawer LL, Moore FA. Persistent inflammation and immunosuppression: a common syndrome and new horizon for surgical intensive care. J Trauma Acute Care Surg. 2012 Jun;72(6):1491-501. doi: 10.1097/TA.0b013e318256e000. PMID 22695412
- [Background] Vanzant EL, Lopez CM, Ozrazgat-Baslanti T, Ungaro R, Davis R, Cuenca AG, Gentile LF, Nacionales DC, Cuenca AL, Bihorac A, Leeuwenburgh C, Lanz J, Baker HV, McKinley B, Moldawer LL, Moore FA, Efron PA. Persistent inflammation, immunosuppression, and catabolism syndrome after severe blunt trauma. J Trauma Acute Care Surg. 2014 Jan;76(1):21-9; discussion 29-30. doi: 10.1097/TA.0b013e3182ab1ab5. PMID 24368353
- [Background] Ellis N, Hughes C, Mazurak V, Joynt C, Larsen B. Does Persistent Inflammatory Catabolic Syndrome Exist in Critically Ill Neonates? JPEN J Parenter Enteral Nutr. 2017 Nov;41(8):1393-1398. doi: 10.1177/0148607116672621. Epub 2016 Oct 10. PMID 27875283